CLINICAL TRIAL: NCT00952029
Title: Multicenter Phase III Randomized Study of FOLFIRI Plus Bevacizumab Following or Not by a Maintenance Therapy With Bevacizumab in Patients With Non-Pretreated Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy and Bevacizumab With or Without Bevacizumab Maintenance Therapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 9; FFCD-PRODIGE-9; FFCD-0802; EU-20912; EU-21030; EUDRACT-2008-007928-25; EUDRACT-2009-017996-11
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance with bevacizumab (Experimental): FOLFIRI + Avastin and during the chemotherapy-free interval maintenance with bevacizumab
  Interventions: Biological: bevacizumab; Drug: FOLFIRI regimen; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium
- No maintenance with bevacizumab (Active Comparator): FOLFIRI + Avastin and during the chemotherapy-free interval NO maintenance
  Interventions: Biological: bevacizumab; Drug: FOLFIRI regimen; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: bevacizumab
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bevacizumab may stop the growth of colorectal cancer by blocking blood flow to the tumor. It is not yet known whether giving more than one drug (combination chemotherapy) is more effective when given with or without bevacizumab in treating patients with metastatic colorectal cancer.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy with or without bevacizumab to see how well it works in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-control duration in patients with metastatic colorectal cancer receiving FOLFIRI chemotherapy in combination with bevacizumab with or without bevacizumab maintenance therapy.

Secondary

* Determine objective response rate.
* Determine non-hematologic grade 3-4 (except alopecia) toxicity rate.
* Determine overall toxicity rate.
* Determine duration of chemotherapy-free interval.
* Determine progression-free survival.
* Determine overall survival.
* Determine time-to-treatment failure.
* Determine quality of life (EORTC QLQ-C30).
* Complete geriatric evaluation.

OUTLINE: This is a multicenter study. Patients are stratified according to cancer center, primary tumor (resected vs unresected), and Köhne criteria (low vs intermediate vs high). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1-2. Chemotherapy treatment repeats every 2 weeks for 12 courses. Patients also receive bevacizumab IV over 30-90 minutes once every 2 weeks during chemotherapy. Patients then receive bevacizumab maintenance therapy once every 2 weeks during the chemotherapy-free interval.
* Arm B: Patients receive FOLFIRI chemotherapy and bevacizumab as in arm A. Patients receive no treatment during the chemotherapy-free interval.

In all arms, the chemotherapy treatment and the chemotherapy-free interval treatment repeats in the absence of disease progression during the chemotherapy portion or unacceptable toxicity. Patients who progress during the chemotherapy-free interval will receive 12 more courses of chemotherapy.

All patients complete quality of life questionnaires (QLQ-30) and patients ≥ 75 also complete the geriatric questionnaire at baseline and every 8 weeks during study treatment.

After completion of study treatment, patients are followed up every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Metastatic disease
* Not a candidate for curative surgery
* At least 1 tumor target measurable by RECIST criteria
* No metastasis potentially resectable after receiving chemotherapy
* No occlusive tumors
* No macronodular peritoneal carcinomatosis
* No known or suspected CNS metastases

PATIENT CHARACTERISTICS:

* OMS status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN in the presence of hepatic metastases)
* Creatinine ≤ 1.5 times ULN
* Proteinuria ≤1 g
* Not pregnant or nursing
* No gastroduodenal ulcer, wound, or fractured bone
* No acute or subacute intestinal occlusion or history of inflammatory bowel disease or large resection of small bowel
* No clinically relevant coronary artery disease or a history of a myocardial infarction within the last 6 months
* No uncontrolled hypertension while receiving chronic medication
* No other malignancy within the past 5 years except for basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* No medical or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study

PRIOR CONCURRENT THERAPY:

* See Patient Characteristics
* No prior chemotherapy for metastatic disease

  * Adjuvant chemotherapy allowed provided it was completed > 6 months ago
* No prior irinotecan or other antiangiogenic therapy
* At least 4 weeks since surgery (except for diagnostic biopsy) or irradiation
* No other drugs not allowed for medical reasons
* Concurrent oral anticoagulants (e.g., coumadin, warfarin) allowed provided the INR is closely monitored

  * A change of anticoagulants to low-molecular weight heparin is preferred

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Disease-control duration | one year after last patient included

SECONDARY OUTCOMES:
Objective response rate | one year after last patient is included
Rate of non-hematologic grade 3-4 toxicities (except alopecia) | one year after last patient is included
Overall toxicity rate | one year after last patient is included
Duration of chemotherapy-free interval | one year after last patient is included
Progression-free survival | one year after last patient is included
Overall survival | one and 2 year after last patient is included
Time-to-treatment failure | one year after last patient is included
Quality of life as assessed by EORTC QLQ-C30 | one year after last patient is included
Geriatric evaluation | one year after last patient is included

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aparicio, Pr, Principal Investigator — Hopital Avicenne BOBIGNY
Locations (102):
- France (102):
  - CH, Abbeville
  - Centre Radiothérapie et Oncologie de Moyenne Garonne, Agen
  - CHU, Amiens
  - Centre Paul Papin, Angers
  - CHU, Angers
  - Pringny, Annecy
  - CH, Aubenas
  - CH, Auxerre
  - Polyclinique Sainte Marguerite, Auxerre
  - CH, Avignon
  - Ch, Bayonne
  - CH, Beauvais
  - CHU, Besançon
  - Centre Pierre Curie, Beuvry
  - CH, Béziers
  - Ch, Blois
  - Hôpital Avicenne, Bobigny
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - CH, Bourg-en-Bresse
  - CH, Bourges
  - CH, Cahors
  - CHIC, Castres
  - Hôpital Privé Sainte Marie, Chalon-sur-Saône
  - CH, Cholet
  - Clinique des Cèdres, Cornebarrieu
  - CH, Créteil
  - CH, Dax
  - Centre Léonard de Vinci, Dechy
  - Centre Leclerc, Dijon
  - CHU, Dijon
  - Parc, Dijon
  - CH, Dunkirk
  - CH, Elbeuf
  - CH, Fréjus
  - Hôpital Chicas, Gap
  - CH, La Roche-sur-Yon
  - CH, Langres
  - CH, Le Mans
  - CH, Libourne
  - Centre Bourgogne, Lille
  - Clinique F. Chenieux, Limoges
  - CH, Longjumeau
  - CHBS, Lorient
  - Centre Léon Bérard, Lyon
  - CHU Edouard Herriot, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Clinique Mutualiste, Lyon
  - Croix Rousse, Lyon
  - Hôpital Saint Joseph, Lyon
  - CHU La Timone, Marseille
  - Hôpital A. Paré, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Saint Joseph, Marseille
  - CH, Mâcon
  - CH, Meaux
  - CHG, Mont-de-Marsan
  - CH, Montauban
  - CH, Montélimar
  - CH Le Raincy, Montfermeil
  - Centre Cancérologique, Montpellier
  - Centre Azuréen, Mougins
  - Hôpital Saint Herblain, Nantes
  - Polyclinique, Narbonne
  - CH, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - L'Archet II, Nice
  - CHU, Nîmes
  - Clinique Valdegour, Centre ONCOGARD - Institut de Cancérologie du Gard, Nîmes
  - CHR (Oncologie Médicale), Orléans
  - CHR, Orléans
  - Clinique Les Murlins, Orléans
  - Bichat, Paris
  - CHU - Kremlin Bicêtre, Paris
  - HEGP, Paris
  - Hôpital Saint Louis, Paris
  - Pitié Salpetière, Paris
  - CH, Pau
  - CH, Perpignan
  - CH, Pessac
  - CH, Périgueux
  - CH, Rang-du-Fliers
  - CH, Reims
  - CH, Romans-sur-Isère
  - CH, Roubaix
  - CHU, Rouen
  - CH, Saint-Brieuc
  - Clinique Armoricaine, Saint-Brieuc
  - HIA Begin, Saint-Mandé
  - Centre Joliot Curie, Saint-Martin-Boulogne
  - Clinique Mutualiste, Saint-Nazaire
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - CHU Trousseau, Tours
  - CH, Valence
  - Clinique Générale, Valence
  - CH, Valenciennes
  - CAC, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - Clinique, Vienne
  - CH, Villejuif
  - Hôpital Intercommunal, Villeneuve-Saint-Georges

REFERENCES:
- [Background] Aparicio T, Linot B, Le Malicot K, Bouche O, Boige V, Francois E, Ghiringhelli F, Legoux JL, Ben Abdelghani M, Phelip JM, Faroux R, Dahan L, Taieb J, Bedenne L. FOLFIRI+bevacizumab induction chemotherapy followed by bevacizumab or observation in metastatic colorectal cancer, a phase III trial (PRODIGE 9--FFCD 0802). Dig Liver Dis. 2015 Apr;47(4):271-2. doi: 10.1016/j.dld.2015.01.146. Epub 2015 Jan 20. No abstract available. PMID 25677925
- [Result] Aparicio T, Ghiringhelli F, Boige V, Le Malicot K, Taieb J, Bouche O, Phelip JM, Francois E, Borel C, Faroux R, Dahan L, Jacquot S, Genet D, Khemissa F, Suc E, Desseigne F, Texereau P, Lepage C, Bennouna J; PRODIGE 9 Investigators. Bevacizumab Maintenance Versus No Maintenance During Chemotherapy-Free Intervals in Metastatic Colorectal Cancer: A Randomized Phase III Trial (PRODIGE 9). J Clin Oncol. 2018 Mar 1;36(7):674-681. doi: 10.1200/JCO.2017.75.2931. Epub 2018 Jan 18. PMID 29346040
- [Result] Aparicio T, Bennouna J, Le Malicot K, Boige V, Taieb J, Bouche O, Phelip JM, Francois E, Borel C, Faroux R, Dahan L, Bachet JB, Egreteau J, Kaminsky MC, Gornet JM, Cojocarasu O, Gasmi M, Guerin-Meyer V, Lepage C, Ghiringhelli F; for PRODIGE investigators/collaborators. Predictive factors for early progression during induction chemotherapy and chemotherapy-free interval: analysis from PRODIGE 9 trial. Br J Cancer. 2020 Mar;122(7):957-962. doi: 10.1038/s41416-020-0735-8. Epub 2020 Feb 4. PMID 32015513
- [Derived] Guilloteau A, Abrahamowicz M, Boussari O, Jooste V, Aparicio T, Quantin C, Le Malicot K, Binquet C. Impact of time-varying cumulative bevacizumab exposures on survival: re-analysis of data from randomized clinical trial in patients with metastatic colo-rectal cancer. BMC Med Res Methodol. 2021 Jan 9;21(1):14. doi: 10.1186/s12874-020-01202-9. PMID 33422006
- [Derived] Dohan A, Gallix B, Guiu B, Le Malicot K, Reinhold C, Soyer P, Bennouna J, Ghiringhelli F, Barbier E, Boige V, Taieb J, Bouche O, Francois E, Phelip JM, Borel C, Faroux R, Seitz JF, Jacquot S, Ben Abdelghani M, Khemissa-Akouz F, Genet D, Jouve JL, Rinaldi Y, Desseigne F, Texereau P, Suc E, Lepage C, Aparicio T, Hoeffel C; PRODIGE 9 Investigators and PRODIGE 20 Investigators. Early evaluation using a radiomic signature of unresectable hepatic metastases to predict outcome in patients with colorectal cancer treated with FOLFIRI and bevacizumab. Gut. 2020 Mar;69(3):531-539. doi: 10.1136/gutjnl-2018-316407. Epub 2019 May 17. PMID 31101691